CLINICAL TRIAL: NCT01668784
Title: A Randomized, Open-Label, Phase 3 Study of Nivolumab (BMS-936558) vs. Everolimus in Subjects With Advanced or Metastatic Clear-Cell Renal Cell Carcinoma Who Have Received Prior Anti-Angiogenic Therapy
Brief Title: Study of Nivolumab (BMS-936558) vs. Everolimus in Pre-Treated Advanced or Metastatic Clear-cell Renal Cell Carcinoma (CheckMate 025)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA209-025; 2011-005132-26 (EudraCT Number)
Expanded Access: NCT03126643 (Approved for marketing)
Record Dates: First submitted 2012-08-16; First posted 2012-08-20 (Estimated); Results first posted 2016-04-29 (Estimated); Last update posted 2022-08-09 (Actual); Status verified 2022-07

CONDITIONS: Advanced or Metastatic (Medically or Surgically Unresectable) Clear-cell Renal Cell Carcinoma
MeSH Terms: conditions — Neoplasm Metastasis; Carcinoma, Renal Cell | interventions — Nivolumab; Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1: Nivolumab (Experimental): Nivolumab 3 mg/kg solution intravenously every 2 weeks until documented disease progression, discontinuation due to toxicity, withdrawal of consent or the study ends
  Interventions: Biological: Nivolumab
- Arm 2: Everolimus (Active Comparator): Everolimus 10 mg tablets by mouth daily until documented disease progression, discontinuation due to toxicity, withdrawal of consent or the study ends
  Interventions: Drug: Everolimus

INTERVENTIONS:
Biological: Nivolumab
  Other Names: BMS-936558
  Arms: Arm 1: Nivolumab
Drug: Everolimus
  Other Names: Afinitor
  Arms: Arm 2: Everolimus

SUMMARY:
The purpose of the study is to compare the clinical benefit, as measured by duration of overall survival, of Nivolumab vs. Everolimus in subjects with advanced or metastatic clear-cell renal cell carcinoma who have received prior anti-angiogenic therapy

ELIGIBILITY:
Inclusion Criteria:

* Men & women ≥18 years of age
* Histologic confirmation of renal cell carcinoma (RCC) with clear-cell component
* Advanced/metastatic RCC
* Measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria
* Received 1 or 2 prior anti-angiogenic therapy regimens in advanced or metastatic setting
* No more than 3 total prior systemic treatment regimens in the advanced or metastatic setting, and evidence of progression on or after last treatment regimen received and within 6 months of enrollment
* Karnofsky Performance Score ≥70%

Exclusion Criteria:

* Any Central Nervous System (CNS) metastases or history of CNS metastases
* Prior therapy with an Mammalian target of rapamycin (mTOR) inhibitor
* Any active known or suspected autoimmune disease
* Uncontrolled adrenal insufficiency
* Active chronic liver disease
* Prior malignancy active within past 3 years, except for locally curable cancers

Other protocol-defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 821 (Actual)
Dates: Start 2012-10-09 (Actual); Primary Completion 2015-05-06 (Actual); Study Completion 2021-07-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (154):
- United States (39):
  - Local Institution - 0182, Fayetteville, Arkansas
  - UCSD Moores Cancer Center, La Jolla, California
  - Local Institution - 0024, Los Angeles, California
  - University Of Southern California, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Ucsf Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Stanford Cancer Institute, Stanford, California
  - University Of Colorado, Aurora, Colorado
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Local Institution - 0027, Washington D.C., District of Columbia
  - H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida
  - Winship Cancer Institute., Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Loyola University Chicago, Maywood, Illinois
  - Indiana University Simon Cancer Center, Indianapolis, Indiana
  - University Of Iowa Hospitals And Clinics, Iowa City, Iowa
  - Sidney Kimmel Comprehensive Cancer Center At Johns Hopkins, Baltimore, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University Of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Karmanos Cancer Institute, Detroit, Michigan
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Roswell Park Cancer Institute, Buffalo, New York
  - Memorial Sloan Kettering Nassau, New York, New York
  - Weill Cornell Medical College, New York, New York
  - Levine Cancer Institute, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - The Ohio State University, Columbus, Ohio
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Medical University Of South Carolina, Charleston, South Carolina
  - St Francis Hospital, Greenville, South Carolina
  - Tennessee Oncology, PLLC, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Ut Southwestern Medical Center, Dallas, Texas
  - Local Institution - 0139, Houston, Texas
  - CTRC at UTHSC San Antonio, San Antonio, Texas
  - Local Institution - 0076, Richmond, Virginia
  - Local Institution - 0009, Seattle, Washington
  - University Of Washington, Seattle, Washington
- Argentina (5):
  - COIBA, Berazategui, Buenos Aires
  - Local Institution, Capital Federal, Buenos Aires
  - Centro Para La Atencion Integral Del Paciente Oncologico, San Miguel de Tucumán, Tucumán Province
  - Local Institution, Buenos Aires
  - Instituto Oncologico De Cordoba, Córdoba
- Australia (5):
  - Local Institution - 0095, Westmead, New South Wales
  - Local Institution, Woodville South, South Australia
  - Local Institution, Box Hill, Victoria
  - Local Institution, Clayton, Victoria
  - Local Institution, Melbourne, Victoria
- Austria (2):
  - Local Institution, Linz
  - Local Institution, Vienna
- Belgium (3):
  - Local Institution, Brussels
  - Local Institution, Ghent
  - Local Institution, Leuven
- Brazil (3):
  - Local Institution - 0125, Ijuí, Rio Grande do Sul
  - Local Institution - 0124, São Paulo
  - Local Institution, São Paulo
- Canada (9):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - BC Cancer Agency - Vancouver Centre, Vancouver, British Columbia
  - Centre D'Oncologie Dr-Leon-Richard, Moncton, New Brunswick
  - QEII Health Sciences Centre, Halfax, Nova Scotia
  - Local Institution - 0143, Oshawa, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - Chum, Hopital Notre-Dame, Montreal, Quebec
  - Local Institution - 0145, Montreal
- Czechia (3):
  - Local Institution, Hradec Králové
  - Local Institution, Olomouc
  - Local Institution, Prague
- Denmark (3):
  - Local Institution, Aarhus N
  - Local Institution, Herlev
  - Local Institution - 0137, Odense
- Local Institution, Helsinki, Finland
- France (17):
  - Local Institution - 0006, Vandœuvre-lès-Nancy, Lorraine
  - Local Institution - 0008, Bordeaux
  - Local Institution, Bordeaux
  - Local Institution - 0007, Lyon
  - Local Institution, Lyon
  - Local Institution - 0004, Marseille
  - Local Institution, Marseille
  - Local Institution - 0118, Paris
  - Local Institution - 0003, Poitiers
  - Local Institution, Poitiers
  - Local Institution - 0005, Saint-Herblain
  - Local Institution, Saint-Herblain
  - Local Institution - 0012, Toulouse
  - Local Institution, Toulouse
  - Local Institution, Vandœuvre-lès-Nancy
  - Local Institution - 0002, Villejuif
  - Local Institution, Villejuif
- Germany (8):
  - Local Institution, Aachen
  - Local Institution, Dresden
  - Local Institution, Erlangen
  - Local Institution, Essen
  - Local Institution, Hanover
  - Local Institution - 0126, Heidelberg
  - Local Institution, Munich
  - Local Institution, Tübingen
- Greece (2):
  - Alexandra General Hospital Of Athens, Athens
  - Euromedica General Clinic of Thessaloniki, Thessaloniki
- Ireland (3):
  - Local Institution, Tallaght, Dublin
  - Local Institution - 0087, Dublin
  - Local Institution, Dublin
- Israel (4):
  - Local Institution, Haifa
  - Local Institution - 0148, Petah Tikva
  - Local Institution, Ramat Gan
  - Local Institution, Tel Aviv
- Italy (8):
  - Local Institution, Arezzo
  - Local Institution, Meldola (fc)
  - Local Institution - 0082, Milan
  - Local Institution, Rimini
  - Local Institution, Roma
  - Local Institution - 0102, Rozzano
  - Local Institution, Siena
  - Local Institution, Terni
- Japan (15):
  - Local Institution, Akita, Akita
  - Local Institution, Chiba, Chiba
  - Local Institution, Higashiku, Fukuoka
  - Local Institution, Sapporo, Hokkaido
  - Local Institution, Morioka, Iwate
  - Local Institution, Yokohama, Kanagawa
  - Local Institution, Kyoto, Kyoto
  - Local Institution, Osaka-sayama-shi, Osaka
  - Local Institution - 0169, Suita, Osaka
  - Local Institution - 0167, Hamamatsu, Shizuoka
  - Local Institution, Tokushima, Tokushima
  - Local Institution, Yamagata, Yamagata
  - Local Institution, Kobe-city, Hyogo
  - Local Institution, Kumamoto
  - Local Institution, Tokyo
- Norway (2):
  - Local Institution, Bergen
  - Local Institution, Lorenskog
- Poland (6):
  - Local Institution, Gdansk
  - Local Institution, Lodz
  - Local Institution, Poznan
  - Local Institution, Rybnik
  - Local Institution, Warsaw
  - Local Institution, Wroclaw
- Romania (4):
  - Local Institution, Bucharest
  - Local Institution, Craiova
  - Local Institution, Iași
  - Local Institution, Timișoara
- Russia (2):
  - Local Institution, Moscow
  - Local Institution, Saint Petersburg
- Spain (4):
  - Local Institution, Pamplona, Navarre
  - Local Institution, Barcelona
  - Local Institution - 0064, L'Hospitalet de Llobregat
  - Local Institution, Madrid
- Sweden (2):
  - Local Institution, Gothenberg
  - Local Institution, Solna
- United Kingdom (4):
  - Local Institution, Cambridge, Cambridgeshire
  - Local Institution - 0048, Swansea, Carmarthenshire
  - Local Institution, Swansea, Carmarthenshire
  - Local Institution, London, Greater London

REFERENCES:
- [Derived] Klijn SL, Fenwick E, Kroep S, Johannesen K, Malcolm B, Kurt M, Kiff C, Borrill J. What Did Time Tell Us? A Comparison and Retrospective Validation of Different Survival Extrapolation Methods for Immuno-Oncologic Therapy in Advanced or Metastatic Renal Cell Carcinoma. Pharmacoeconomics. 2021 Mar;39(3):345-356. doi: 10.1007/s40273-020-00989-1. Epub 2021 Jan 11. PMID 33428174
- [Derived] Ambavane A, Yang S, Atkins MB, Rao S, Shah A, Regan MM, McDermott DF, Michaelson MD. Clinical and economic outcomes of treatment sequences for intermediate- to poor-risk advanced renal cell carcinoma. Immunotherapy. 2020 Jan;12(1):37-51. doi: 10.2217/imt-2019-0199. Epub 2020 Jan 29. PMID 31992108
- [Derived] Shah R, Botteman M, Solem CT, Luo L, Doan J, Cella D, Motzer RJ. A Quality-adjusted Time Without Symptoms or Toxicity (Q-TWiST) Analysis of Nivolumab Versus Everolimus in Advanced Renal Cell Carcinoma (aRCC). Clin Genitourin Cancer. 2019 Oct;17(5):356-365.e1. doi: 10.1016/j.clgc.2019.05.010. Epub 2019 May 31. PMID 31272883
- [Derived] Long GV, Tykodi SS, Schneider JG, Garbe C, Gravis G, Rashford M, Agrawal S, Grigoryeva E, Bello A, Roy A, Rollin L, Zhao X. Assessment of nivolumab exposure and clinical safety of 480 mg every 4 weeks flat-dosing schedule in patients with cancer. Ann Oncol. 2018 Nov 1;29(11):2208-2213. doi: 10.1093/annonc/mdy408. PMID 30215677
- [Derived] Escudier B, Motzer RJ, Sharma P, Wagstaff J, Plimack ER, Hammers HJ, Donskov F, Gurney H, Sosman JA, Zalewski PG, Harmenberg U, McDermott DF, Choueiri TK, Richardet M, Tomita Y, Ravaud A, Doan J, Zhao H, Hardy H, George S. Treatment Beyond Progression in Patients with Advanced Renal Cell Carcinoma Treated with Nivolumab in CheckMate 025. Eur Urol. 2017 Sep;72(3):368-376. doi: 10.1016/j.eururo.2017.03.037. Epub 2017 Apr 12. PMID 28410865
- [Derived] Escudier B, Sharma P, McDermott DF, George S, Hammers HJ, Srinivas S, Tykodi SS, Sosman JA, Procopio G, Plimack ER, Castellano D, Gurney H, Donskov F, Peltola K, Wagstaff J, Gauler TC, Ueda T, Zhao H, Waxman IM, Motzer RJ; CheckMate 025 investigators. CheckMate 025 Randomized Phase 3 Study: Outcomes by Key Baseline Factors and Prior Therapy for Nivolumab Versus Everolimus in Advanced Renal Cell Carcinoma. Eur Urol. 2017 Dec;72(6):962-971. doi: 10.1016/j.eururo.2017.02.010. Epub 2017 Mar 3. PMID 28262413
- [Derived] Cella D, Grunwald V, Nathan P, Doan J, Dastani H, Taylor F, Bennett B, DeRosa M, Berry S, Broglio K, Berghorn E, Motzer RJ. Quality of life in patients with advanced renal cell carcinoma given nivolumab versus everolimus in CheckMate 025: a randomised, open-label, phase 3 trial. Lancet Oncol. 2016 Jul;17(7):994-1003. doi: 10.1016/S1470-2045(16)30125-5. Epub 2016 Jun 6. PMID 27283863
- [Derived] Motzer RJ, Escudier B, McDermott DF, George S, Hammers HJ, Srinivas S, Tykodi SS, Sosman JA, Procopio G, Plimack ER, Castellano D, Choueiri TK, Gurney H, Donskov F, Bono P, Wagstaff J, Gauler TC, Ueda T, Tomita Y, Schutz FA, Kollmannsberger C, Larkin J, Ravaud A, Simon JS, Xu LA, Waxman IM, Sharma P; CheckMate 025 Investigators. Nivolumab versus Everolimus in Advanced Renal-Cell Carcinoma. N Engl J Med. 2015 Nov 5;373(19):1803-13. doi: 10.1056/NEJMoa1510665. Epub 2015 Sep 25. PMID 26406148
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 803 Participants Treated
Groups:
- Nivolumab: Nivolumab at 3 mg/kg solution provided intravenously every 2 weeks until documented disease progression, discontinuation due to toxicity, withdrawal of consent or the study ends.
- Everolimus: Everolimus provided in 10 mg tablets by mouth daily until documented disease progression, discontinuation due to toxicity, withdrawal of consent or the study ends.
Period: Randomized (Pre-treatment)
Arm/Group | Nivolumab | Everolimus
Started | 410 | 411
Completed | 406 | 397
Not Completed | 4 | 14
Not completed — Disease Progression | 0 | 1
Not completed — Request to Discontinue Study Treatment | 0 | 3
Not completed — Withdrawal by Subject | 1 | 8
Not completed — Poor/Non-Compliance | 1 | 0
Not completed — No Longer Meets Study Criteria | 2 | 1
Not completed — participant requested to be treated a local facility | 0 | 1
Period: Treatment Period
Arm/Group | Nivolumab | Everolimus
Started | 406 | 397
Completed | 0 | 0
Not Completed | 406 | 397
Not completed — Disease Progression | 316 | 293
Not completed — Study Drug Toxicity | 46 | 53
Not completed — Death | 1 | 1
Not completed — Adverse Event Unrelated to Study Drug | 14 | 14
Not completed — Request to Discontinue Study Treatment | 14 | 21
Not completed — Withdrawal by Subject | 5 | 3
Not completed — Maximal Clinical Benefit | 3 | 3
Not completed — Other | 2 | 8
Not completed — Administrative Reason by Sponsor | 5 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants; any participant that was randomized to any treatment group in the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Nivolumab | Everolimus | Total
Number analyzed (Participants) | 410 | 411 | 821
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.6 (10.87) | 61.9 (10.43) | 61.3 (10.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 95 | 107 | 202
  Male | 315 | 304 | 619
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 42 | 32 | 74
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 1 | 4 | 5
  White | 353 | 367 | 720
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 13 | 7 | 20

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS) at Primary Endpoint
Description: Overall Survival (OS) was defined as the time from randomization to the date of death. Participants that had not died were censored at last known date alive. Median OS time was calculated using Kaplan-Meier Estimates. Interim analysis for the Primary Endpoint occurred after 398 deaths (70% of the total OS events needed for final analysis). At that time the data monitoring committee noted that the pre-specified boundary for OS (nominal significance level p < 0.0148) was crossed while no new safety signals that would affect continuation of the study were found. The study was stopped early by the Sponsor, Bristol-Myers Squibb (BMS) and the interim analysis became the final analysis. As a result, participants in the everolimus groups could be assessed for a crossover to nivolumab treatment if they met all inclusion criteria.
Time Frame: Randomization until 398 deaths, up to May 2015 (approximately 30 months)
Population: All randomized participants; any participants that was randomized to any treatment group in the study.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nivolumab | Everolimus
Number analyzed (Participants) | 410 | 411
months | 25.00 [21.75 to NA] — N.A.: Not Available: Too few events to estimate the upper limit of the confidence interval | 19.55 [17.64 to 23.06]
Statistical Analysis 1: Comparison: Nivolumab vs Everolimus; Test type: Superiority; p = 0.0018, Log Rank — The boundary for statistical significance required the p-value to be less than 0.0148 at the interim analyses; Log-rank Test stratified by the Memorial Sloan-Kettering Cancer Center risk group, number of prior anti-angiogenic therapies, and the region; Hazard Ratio (HR) = 0.73, 98.52% CI 2-sided [0.57 to 0.93] — Stratified Cox proportional hazard model. Hazard ratio (HR) was Nivolumab over Everolimus

2. Secondary Outcome: Investigator-assessed Objective Response Rate (ORR)
Description: ORR is defined as Percentage of participants with a best response of complete response (CR) or partial response (PR) divided by number of randomized participants. CR=Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm.; PR=At least a 30% decrease in the sum of diameters of target lesions, the baseline sum diameters used as reference. Tumor assessments began at 8 weeks following randomization and continued every 8 weeks for the first year, then every 12 weeks thereafter until disease progression or death. CIs used Clopper and Pearson.
Time Frame: from randomization up to disease progression or death (approximately up to 105 Months)
Population: All randomized participants; any participants that was randomized to any treatment group in the study.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Nivolumab | Everolimus
Number analyzed (Participants) | 410 | 411
percentage of participants | 25.9 [21.7 to 30.4] | 6.1 [4.0 to 8.8]

3. Secondary Outcome: Investigator-assessed Duration of Objective Response
Description: Duration of objective response is defined as the time from study start date to response, CR or partial response, PR) to the date of the first documented tumor progression as determined by the investigator (per RECIST 1.1 criteria or clinical) or death due to any cause, whichever occurred first. For participants who neither progress nor die, the duration of objective response were censored at the same time they were censored for the primary definition. CR=Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm.; PR=At least a 30% decrease in the sum of diameters of target lesions, the baseline sum diameters used as reference. Based on Kaplan-Meier Estimates.
Time Frame: From randomization to date of disease progression or death or censoring if no progression or death occurred (approximately 105 months)
Population: All randomized participants with a response; any participants that were randomized to any treatment group in the study and that had a response.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nivolumab | Everolimus
Number analyzed (Participants) | 106 | 25
months | 13.11 [9.26 to 19.75] | 10.18 [5.39 to 18.73]

4. Secondary Outcome: Investigator-assessed Time to Objective Response
Description: Time to objective response is defined as the time from randomization to first response (complete response, CR or partial response, PR). CR=Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm.; PR=At least a 30% decrease in the sum of diameters of target lesions, the baseline sum diameters used as reference.
Time Frame: Randomization to date of first response (approximately 105 months)
Population: All randomized participants with a response; any participants that was randomized to any treatment group in the study and that had a response.
Measure: Median (Full Range); unit: months
Arm/Group | Nivolumab | Everolimus
Number analyzed (Participants) | 106 | 25
months | 3.55 [1.4 to 24.8] | 3.71 [1.5 to 68.9]

5. Secondary Outcome: Investigator-assessed Time of Progression-free Survival (PFS)
Description: PFS=time from randomization to date of first documented tumor progression as determined by investigator (per RECIST 1.1 criteria or clinical) or death due to any cause, whichever occurred first. Participants who die without a reported prior progression and without subsequent anti-cancer therapy were considered to have progressed on the date of their death. Participants who did not progress or die were censored on the date of their last evaluable tumor assessment. Participants who did not have any on-study tumor assessments and did not die were censored on the date they were randomized. Participants who received any subsequent anti-cancer therapy without a prior reported progression were censored at the last evaluable tumor assessment prior to or on initiation date of the subsequent anti-cancer therapy. Progressive disease: >=20% increase in sum of target lesion diameters and sum must show absolute increase of >=5mm; smallest sum on study as reference. Based on Kaplan-Meier Estimates.
Time Frame: from randomization up to disease progression or death (approximately up to 105 Months)
Population: All randomized participants; any participants that was randomized to any treatment group in the study.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nivolumab | Everolimus
Number analyzed (Participants) | 410 | 411
months | 4.21 [3.68 to 5.36] | 4.50 [3.71 to 5.52]
Statistical Analysis 1: Comparison: Nivolumab vs Everolimus; Test type: Superiority; p = 0.0340, Log Rank; Log-rank Test stratified by the Memorial Sloan-Kettering Cancer Center (MSKCC) risk group, number of prior anti-angiogenic therapies, and the region; Hazard Ratio (HR) = 0.84, 95% CI 2-sided [0.72 to 0.99] — Stratified Cox proportional hazard model. Hazard ratio is nivolumab over everolimus

6. Secondary Outcome: Overall Survival (OS) by Programmed Death-Ligand 1 (PD-L1) Expression Level
Description: Quantifiable PD-L1 expression=percent of tumor cell membrane staining in a minimum of 100 evaluable tumor cells per Dako PD-L1 IHC assay. If the PD-L1 staining could not be quantified it was classified as: indeterminate=tumor cell membrane staining hampered for reasons attributed to biology of tumor biopsy specimen and not due to improper sample preparation or handling; not evaluable=tumor biopsy specimen was not optimally collected or prepared. Not evaluable determined from H&E process before the tumor biopsy specimen was sent for evaluation or from H&E process during PD-L1 evaluation; baseline PD-L1 expression=if more than one tumor biopsy specimen was available, the most recently collected specimen with a quantifiable result. If all specimens for a given participant are either indeterminate or not evaluable, then the PD-L1 expression was considered indeterminate as long as at least one specimen is indeterminate. Otherwise, PD-L1 expression was considered not evaluable.
Time Frame: Randomization to date of death or date of last contact for patients without documentation of death, up to May 2015 (approximately 30 months)
Population: PD-L1 quantifiable participants; All randomized participants with quantifiable PD-L1 expression at baseline
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nivolumab | Everolimus
Number analyzed (Participants) | 370 | 386
months
  Participant PD-L1 expression >=1%: number analyzed (Participants) | 94 | 87
  Participant PD-L1 expression >=1% | 5.36 [2.04 to 7.46] | 4.17 [3.09 to 5.52]
  Participant PD-L1 expression <1%: number analyzed (Participants) | 276 | 299
  Participant PD-L1 expression <1% | 3.94 [3.68 to 5.36] | 4.67 [3.71 to 5.72]

7. Secondary Outcome: Number of Participants With Serious Adverse Events, Death, Discontinuation Due to Adverse Events
Description: Adverse event (AE) defined: any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that may not have a causal relationship with treatment. Serious adverse event (SAE) defined: a medical event that at any dose results in death, persistent or significant disability/incapacity, or drug dependency/abuse; is life-threatening, an important medical event, or a congenital anomaly/birth defect; or requires or prolongs hospitalization.
Time Frame: Day of first dose to 30 days post study completion (approximately 106 months)
Population: All treated participants; all participants who received at least one dose of nivolumab or everolimus
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab | Everolimus
Number analyzed (Participants) | 406 | 397
Participants
  Deaths | 324 | 342
  SAEs | 211 | 177
  Drug related SAEs | 51 | 55
  Drug related AEs | 327 | 353
  Discontinued due to Drug-related AEs | 40 | 51
  Discontinued due to AEs | 85 | 82
  Adverse Events | 398 | 387

8. Secondary Outcome: Percentage of Participants With Disease-related Symptom Progression (DRSP)
Description: Disease-related symptom progression rate (DRSPR)=a decrease of two points in the Functional Assessment of Cancer Therapy-Kidney Symptom Index - Disease Related Symptoms (FKSI-DRS) questionnaire relative to the participant's baseline FKSI-DRS score with no later increase above this threshold observed during the course of the study. The 9 items of the FKSI-DRS were summarized into a symptom scale ranging in score from 0 to 36, with 0 being the worst possible score and 36 being the best possible score. A single measure reporting a decrease of at least 2 units was considered disease-related symptom progression only if it was the last one available for the participant. In order to consider a questionnaire received as valid, over 50% of the items were to be completed. Calculated by the Clopper-Pearson method for each treatment group.
Time Frame: from randomization up to disease progression or death (approximately up to 105 Months)
Population: All randomized participants; any participants that was randomized to any treatment group in the study.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Nivolumab | Everolimus
Number analyzed (Participants) | 410 | 411
percentage of participants
  Disease-related Symptom Progression Rate (DRSPR) | 44.6 [39.0 to 50.3] | 54.6 [49.2 to 60.0]
  DRSPR Including Death and Investigator Progression | 95.5 [92.6 to 97.5] | 99.4 [97.9 to 99.9]

9. Secondary Outcome: Number of Participants Meeting Marked Laboratory Abnormality Criteria in Specific Liver and Thyroid Tests
Description: Aspartate aminotransferase, AST. Alanine aminotransaminase, ALT. Total bilirubin, tBIL. Thyroid stimulating hormone, TSH. Upper limit of normal (ULN). Units per Liter (U/L). Results reported in International System of Units (SI).
Time Frame: Day 1 to 30 days post study completion (approximately 106 months)
Population: To all treated participants with evaluable measurements
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab | Everolimus
Number analyzed (Participants) | 406 | 397
Participants
  ALT or AST > 3.0*ULN: number analyzed (Participants) | 401 | 377
  ALT or AST > 3.0*ULN | 32 | 15
  ALT or AST > 5.0*ULN: number analyzed (Participants) | 401 | 377
  ALT or AST > 5.0*ULN | 20 | 7
  ALT or AST > 10.0*ULN: number analyzed (Participants) | 401 | 377
  ALT or AST > 10.0*ULN | 9 | 1
  ALT or AST > 20.0*ULN: number analyzed (Participants) | 401 | 377
  ALT or AST > 20.0*ULN | 2 | 0
  Total Bilirubin > 2.0*ULN: number analyzed (Participants) | 401 | 376
  Total Bilirubin > 2.0*ULN | 6 | 2
  ALT or AST>3.0*ULN, tBIL>2.0 ULN, 1day: number analyzed (Participants) | 401 | 376
  ALT or AST>3.0*ULN, tBIL>2.0 ULN, 1day | 3 | 0
  ALT or AST>3.0*ULN, tBIL>2.0 ULN,30day: number analyzed (Participants) | 401 | 376
  ALT or AST>3.0*ULN, tBIL>2.0 ULN,30day | 4 | 1
  TSH > ULN: number analyzed (Participants) | 382 | 361
  TSH > ULN | 159 | 78
  TSH < LLN: number analyzed (Participants) | 382 | 361
  TSH < LLN | 60 | 60

10. Secondary Outcome: Number of Participants With Abnormal Hematology and Serum Chemistry Laboratory Parameters by Worse CTC Grade - SI Units
Description: Common Terminology Criteria (CTC) version 4.0 in International System of Units (SI); Gr 3=Severe, Gr 4= Potentially Life-threatening or disabling. Hematology parameters=Hemoglobin (Gr 3: < 8.0 g/dL), Platelet Count (Gr 3: 25.0 -< 50.0*10^9 c/L; Gr 4: < 25.0*10^9 c/L), Leukocyte Count (Gr 3: 1.0 -< 2.0*10^3 c/µL; Gr4: < 1.0*10^3 c/µL), Absolute Lymphocyte Count (Gr 3: 0.2 -< 0.5*10^3 c/µL; Gr 4: < 0.2*10^3 c/µL), Absolute Neutrophil Count (Gr 3: 0.5 - < 1.0*10^3 c/µL; Gr 4: < 0.5*10^3 c/µL). Liver Function parameters=Alkaline Phosphatase (Gr 3: > 5.0 - 20.0 U/L * ULN; Gr 4: > 20.0 U/L * ULN), AST (Gr 3: > 5.0 - 20.0 U/L * ULN; Gr 4: > 20.0 U/L * ULN), ALT (Gr 3: > 5.0 - 20.0 U/L * ULN; Gr 4: > 20.0 U/L * ULN), tBIL (Gr 3: > 3.0 - 10.0 mg/dL * ULN; Gr 4: > 10.0 mg/dL * ULN). Renal parameter=Creatinine (Grade: Gr3: > 3.0 - 6.0 mg/dL *ULN; Gr4: > 6.0 mg/dL *ULN). Cells per microliter (c/µL). Cells per Liter (c/L). Grams per deciliter (g/dL). Milligrams per deciliter (mg/dL).
Time Frame: Day 1 to 30 days post study completion (approximately 106 months)
Population: To all treated participants with evaluable measurements
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab | Everolimus
Number analyzed (Participants) | 406 | 397
Participants
  Hemoglobin, Grade 3: number analyzed (Participants) | 395 | 383
  Hemoglobin, Grade 3 | 33 | 61
  Platelet Count, Grade 3: number analyzed (Participants) | 391 | 379
  Platelet Count, Grade 3 | 1 | 6
  Platelet Count, Grade 4: number analyzed (Participants) | 391 | 379
  Platelet Count, Grade 4 | 0 | 1
  Leukocytes, Grade 3: number analyzed (Participants) | 394 | 380
  Leukocytes, Grade 3 | 0 | 1
  Leukocytes, Grade 4: number analyzed (Participants) | 394 | 380
  Leukocytes, Grade 4 | 1 | 0
  Lymphocytes (absolute), Grade 3: number analyzed (Participants) | 391 | 377
  Lymphocytes (absolute), Grade 3 | 28 | 43
  Lymphocytes (absolute), Grade 4: number analyzed (Participants) | 391 | 377
  Lymphocytes (absolute), Grade 4 | 3 | 6
  Absolute Neutrophil Count, Grade 3: number analyzed (Participants) | 392 | 378
  Absolute Neutrophil Count, Grade 3 | 0 | 2
  Absolute Neutrophil Count, Grade 4: number analyzed (Participants) | 392 | 378
  Absolute Neutrophil Count, Grade 4 | 0 | 1
  Alkaline Phosphatase, Grade 3: number analyzed (Participants) | 400 | 374
  Alkaline Phosphatase, Grade 3 | 11 | 3
  Aspartate Aminotransferase, Grade 3: number analyzed (Participants) | 400 | 375
  Aspartate Aminotransferase, Grade 3 | 9 | 6
  Aspartate Aminotransferase, Grade 4: number analyzed (Participants) | 400 | 375
  Aspartate Aminotransferase, Grade 4 | 2 | 0
  Alanine Aminotransferase, Grade 3: number analyzed (Participants) | 401 | 376
  Alanine Aminotransferase, Grade 3 | 12 | 3
  Alanine Aminotransferase, Grade 4: number analyzed (Participants) | 401 | 376
  Alanine Aminotransferase, Grade 4 | 1 | 0
  Bilirubin Total, Grade 3: number analyzed (Participants) | 401 | 376
  Bilirubin Total, Grade 3 | 3 | 2
  Creatinine, Grade 3: number analyzed (Participants) | 398 | 379
  Creatinine, Grade 3 | 5 | 5
  Creatinine, Grade 4: number analyzed (Participants) | 398 | 379
  Creatinine, Grade 4 | 3 | 1
  Hypercalcemia, Grade 3: number analyzed (Participants) | 339 | 315
  Hypercalcemia, Grade 3 | 7 | 1
  Hypercalcemia, Grade 4: number analyzed (Participants) | 339 | 315
  Hypercalcemia, Grade 4 | 4 | 1
  Hypocalcemia, Grade 3: number analyzed (Participants) | 339 | 315
  Hypocalcemia, Grade 3 | 2 | 4
  Hypocalcemia, Grade 4: number analyzed (Participants) | 339 | 315
  Hypocalcemia, Grade 4 | 1 | 0
  Hyperkalemia, Grade 3: number analyzed (Participants) | 352 | 332
  Hyperkalemia, Grade 3 | 11 | 7
  Hyperkalemia, Grade 4: number analyzed (Participants) | 352 | 332
  Hyperkalemia, Grade 4 | 3 | 0
  Hypokalemia, Grade 3: number analyzed (Participants) | 352 | 332
  Hypokalemia, Grade 3 | 5 | 3
  Hypermagnesmia, Grade 3: number analyzed (Participants) | 196 | 174
  Hypermagnesmia, Grade 3 | 3 | 0
  Hypomagnesmia, Grade 3: number analyzed (Participants) | 196 | 174
  Hypomagnesmia, Grade 3 | 1 | 0
  Hyponatremia, Grade 3: number analyzed (Participants) | 353 | 332
  Hyponatremia, Grade 3 | 26 | 22
  Hyponatremia, Grade 4: number analyzed (Participants) | 353 | 332
  Hyponatremia, Grade 4 | 1 | 1

11. Post Hoc Outcome: Extended Collection to Post Hoc Overall Survival (OS)
Description: Overall Survival (OS) was defined as the time from randomization to the date of death. Participants that had not died were censored at last known date alive. Median OS time was calculated using Kaplan-Meier Estimates. Interim analysis for the Primary Endpoint occurred after 398 deaths (70% of the total OS events needed for final analysis). At that time the data monitoring committee noted that the pre-specified boundary for OS (nominal significance level p < 0.0148) was crossed while no new safety signals that would affect continuation of the study were found. The study was stopped early by the Sponsor, Bristol-Myers Squibb (BMS) and the interim analysis became the final analysis. As a result, participants in the everolimus groups could be assessed for a crossover to nivolumab treatment if they met all inclusion criteria.
  This outcome measure represents an updated version of the primary endpoint to include additional data collection that has occurred after the primary completion date.
Time Frame: from randomization up to disease progression or death (approximately up to 105 months)
Population: All Randomized Participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Nivolumab | Everolimus
Number analyzed (Participants) | 410 | 411
Months | 25.82 [22.21 to 29.77] | 19.55 [17.64 to 21.88]
Statistical Analysis 1: Comparison: Nivolumab vs Everolimus; Test type: Superiority; p = 0.0001, Log Rank; Stratified Cox Proportional hazard Model = 0.74, 95% CI 2-sided [0.63 to 0.86]

ADVERSE EVENTS:
Time Frame: All-cause mortality was assessed from first dose to study completion (up to 105 months). SAEs and Other AEs were assessed from first dose to 100 days following last dose (approximately up to 107 months)
Arm/Group | NIVOLUMAB | EVEROLIMUS
All-Cause Mortality (participants affected / at risk) | 324/406 | 342/397
Serious Adverse Events (participants affected / at risk) | 248/406 | 243/397
Other Adverse Events (participants affected / at risk) | 392/406 | 379/397
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NIVOLUMAB (N=406) | EVEROLIMUS (N=397)
Anaemia (Blood and lymphatic system disorders) | 9 | 15
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Methaemoglobinaemia (Blood and lymphatic system disorders) | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 3 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 1
Angina pectoris (Cardiac disorders) | 3 | 0
Arrhythmia (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 2 | 3
Atrial flutter (Cardiac disorders) | 1 | 1
Atrioventricular block (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 4 | 1
Cardiac failure chronic (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 3
Cardiac ventricular thrombosis (Cardiac disorders) | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0
Left ventricular dysfunction (Cardiac disorders) | 1 | 1
Myocardial infarction (Cardiac disorders) | 7 | 2
Pericardial effusion (Cardiac disorders) | 0 | 2
Supraventricular tachycardia (Cardiac disorders) | 0 | 1
Pancreas divisum (Congenital, familial and genetic disorders) | 1 | 0
Tympanic membrane perforation (Ear and labyrinth disorders) | 1 | 0
Adrenal insufficiency (Endocrine disorders) | 3 | 1
Hypercalcaemia of malignancy (Endocrine disorders) | 1 | 0
Hypopituitarism (Endocrine disorders) | 1 | 0
Corneal disorder (Eye disorders) | 1 | 0
Retinal detachment (Eye disorders) | 0 | 1
Visual impairment (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 5 | 4
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 1 | 3
Autoimmune colitis (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 3 | 0
Constipation (Gastrointestinal disorders) | 5 | 2
Diabetic gastroparesis (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 8 | 3
Enterocolitis (Gastrointestinal disorders) | 1 | 1
Food poisoning (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Haemoperitoneum (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 1 | 0
Immune-mediated enterocolitis (Gastrointestinal disorders) | 0 | 1
Intestinal ischaemia (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 1 | 1
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 0 | 1
Large intestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Large intestine perforation (Gastrointestinal disorders) | 2 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Melaena (Gastrointestinal disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 3 | 2
Oesophageal obstruction (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 2 | 0
Pneumoperitoneum (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 2 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 6
Small intestinal perforation (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 1
Umbilical hernia (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 3 | 0
Asthenia (General disorders) | 1 | 0
Chest pain (General disorders) | 1 | 0
Chills (General disorders) | 0 | 1
Disease progression (General disorders) | 1 | 2
Fatigue (General disorders) | 2 | 3
Gait disturbance (General disorders) | 1 | 0
General physical health deterioration (General disorders) | 4 | 5
Hernia (General disorders) | 0 | 1
Hernia pain (General disorders) | 0 | 1
Hyperpyrexia (General disorders) | 1 | 0
Inadequate analgesia (General disorders) | 2 | 0
Influenza like illness (General disorders) | 1 | 0
Multiple organ dysfunction syndrome (General disorders) | 1 | 1
Non-cardiac chest pain (General disorders) | 2 | 2
Oedema peripheral (General disorders) | 2 | 2
Pain (General disorders) | 4 | 3
Performance status decreased (General disorders) | 0 | 1
Peripheral swelling (General disorders) | 1 | 0
Polyp (General disorders) | 0 | 1
Pyrexia (General disorders) | 7 | 6
Systemic inflammatory response syndrome (General disorders) | 1 | 0
Biliary colic (Hepatobiliary disorders) | 1 | 1
Biliary obstruction (Hepatobiliary disorders) | 0 | 2
Cholecystitis (Hepatobiliary disorders) | 1 | 1
Hepatic cytolysis (Hepatobiliary disorders) | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0
Hepatic pain (Hepatobiliary disorders) | 1 | 0
Hepatitis acute (Hepatobiliary disorders) | 1 | 1
Hepatorenal failure (Hepatobiliary disorders) | 1 | 0
Immune-mediated hepatitis (Hepatobiliary disorders) | 1 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 1 | 0
Anaphylactic reaction (Immune system disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 1
Abdominal infection (Infections and infestations) | 0 | 1
Anal abscess (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 1
Brain abscess (Infections and infestations) | 1 | 0
Bronchiolitis (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 2 | 0
Cellulitis (Infections and infestations) | 2 | 2
Cystitis (Infections and infestations) | 1 | 0
Device related sepsis (Infections and infestations) | 0 | 2
Escherichia infection (Infections and infestations) | 0 | 1
Febrile infection (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 2
Gastroenteritis viral (Infections and infestations) | 1 | 0
Genital infection fungal (Infections and infestations) | 1 | 0
Groin infection (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 1 | 1
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 2 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 2
Lymphangitis (Infections and infestations) | 0 | 1
Meningitis (Infections and infestations) | 0 | 1
Periorbital cellulitis (Infections and infestations) | 1 | 0
Peritonitis bacterial (Infections and infestations) | 0 | 1
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 19 | 25
Pneumonia mycoplasmal (Infections and infestations) | 0 | 1
Psoas abscess (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 9 | 3
Septic shock (Infections and infestations) | 0 | 1
Skin infection (Infections and infestations) | 1 | 1
Soft tissue infection (Infections and infestations) | 1 | 0
Spinal cord infection (Infections and infestations) | 2 | 0
Splenic infection (Infections and infestations) | 0 | 1
Staphylococcal bacteraemia (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 3 | 5
Urosepsis (Infections and infestations) | 4 | 0
Wound infection (Infections and infestations) | 1 | 0
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Clavicle fracture (Injury, poisoning and procedural complications) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 1
Femur fracture (Injury, poisoning and procedural complications) | 1 | 2
Humerus fracture (Injury, poisoning and procedural complications) | 3 | 1
Incision site impaired healing (Injury, poisoning and procedural complications) | 0 | 1
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 1
Post procedural complication (Injury, poisoning and procedural complications) | 1 | 0
Post procedural swelling (Injury, poisoning and procedural complications) | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1
Product administration error (Injury, poisoning and procedural complications) | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 | 0
Wound complication (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 2 | 0
Aspartate aminotransferase increased (Investigations) | 2 | 0
Blood bilirubin increased (Investigations) | 1 | 0
Blood creatinine increased (Investigations) | 2 | 3
Blood culture positive (Investigations) | 1 | 0
Blood glucose increased (Investigations) | 1 | 0
Blood potassium increased (Investigations) | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 1 | 0
General physical condition abnormal (Investigations) | 1 | 2
Haemoglobin decreased (Investigations) | 2 | 0
Lipase increased (Investigations) | 1 | 0
Pancreatic enzymes increased (Investigations) | 0 | 1
Transaminases increased (Investigations) | 1 | 0
Viral test positive (Investigations) | 1 | 0
Cachexia (Metabolism and nutrition disorders) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 3 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 5
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 2
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 1
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 10 | 5
Hyperglycaemia (Metabolism and nutrition disorders) | 5 | 5
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 4
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 2
Back disorder (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 9 | 7
Bone disorder (Musculoskeletal and connective tissue disorders) | 1 | 0
Bone lesion (Musculoskeletal and connective tissue disorders) | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 3 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 3
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Osteitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteolysis (Musculoskeletal and connective tissue disorders) | 2 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 3 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 5 | 4
Soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Acoustic neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Acute lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 0
Duodenal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Intracranial tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lymphangiosis carcinomatosa (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 64 | 85
Metastases to abdominal cavity (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to adrenals (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 | 1
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 3
Metastases to pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to thyroid (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastatic renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 1
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal cell carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Skin cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2
Central nervous system haemorrhage (Nervous system disorders) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 2 | 1
Cerebral ischaemia (Nervous system disorders) | 2 | 0
Cerebrovascular accident (Nervous system disorders) | 3 | 6
Dizziness (Nervous system disorders) | 1 | 0
Dural arteriovenous fistula (Nervous system disorders) | 1 | 0
Encephalopathy (Nervous system disorders) | 1 | 0
Epilepsy (Nervous system disorders) | 0 | 1
Facial spasm (Nervous system disorders) | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 2 | 0
Hyperammonaemic encephalopathy (Nervous system disorders) | 0 | 1
Immune-mediated encephalitis (Nervous system disorders) | 0 | 1
Intracranial pressure increased (Nervous system disorders) | 0 | 1
Intraventricular haemorrhage (Nervous system disorders) | 1 | 0
Memory impairment (Nervous system disorders) | 1 | 0
Nerve compression (Nervous system disorders) | 0 | 1
Nervous system disorder (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 0 | 2
Somnolence (Nervous system disorders) | 1 | 0
Spinal cord compression (Nervous system disorders) | 9 | 1
Syncope (Nervous system disorders) | 2 | 0
Thalamus haemorrhage (Nervous system disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Vasogenic cerebral oedema (Nervous system disorders) | 1 | 0
Device loosening (Product Issues) | 0 | 1
Completed suicide (Psychiatric disorders) | 1 | 1
Confusional state (Psychiatric disorders) | 3 | 1
Delirium (Psychiatric disorders) | 0 | 1
Mental disorder (Psychiatric disorders) | 1 | 0
Mental status changes (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 12 | 6
Dysuria (Renal and urinary disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 3
Nephrolithiasis (Renal and urinary disorders) | 1 | 2
Renal colic (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 7 | 6
Renal impairment (Renal and urinary disorders) | 2 | 1
Renal mass (Renal and urinary disorders) | 1 | 1
Renal tubular necrosis (Renal and urinary disorders) | 0 | 1
Tubulointerstitial nephritis (Renal and urinary disorders) | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 1
Urinary tract obstruction (Renal and urinary disorders) | 2 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 | 8
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 4 | 4
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 16 | 19
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 10 | 13
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 | 8
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pulmonary infarction (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Acute febrile neutrophilic dermatosis (Skin and subcutaneous tissue disorders) | 0 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 2
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0
Aortic dissection (Vascular disorders) | 1 | 0
Circulatory collapse (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 1
Hypertensive crisis (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 3 | 1
Lymphoedema (Vascular disorders) | 0 | 1
Orthostatic hypotension (Vascular disorders) | 1 | 0
Thrombosis (Vascular disorders) | 0 | 1
Venous thrombosis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | NIVOLUMAB (N=406) | EVEROLIMUS (N=397)
Anaemia (Blood and lymphatic system disorders) | 93 | 149
Hypothyroidism (Endocrine disorders) | 39 | 15
Abdominal pain (Gastrointestinal disorders) | 46 | 44
Abdominal pain upper (Gastrointestinal disorders) | 27 | 22
Constipation (Gastrointestinal disorders) | 110 | 93
Diarrhoea (Gastrointestinal disorders) | 122 | 141
Dry mouth (Gastrointestinal disorders) | 30 | 25
Dyspepsia (Gastrointestinal disorders) | 15 | 20
Nausea (Gastrointestinal disorders) | 135 | 139
Stomatitis (Gastrointestinal disorders) | 29 | 125
Vomiting (Gastrointestinal disorders) | 77 | 80
Asthenia (General disorders) | 44 | 71
Chills (General disorders) | 32 | 30
Fatigue (General disorders) | 215 | 196
Malaise (General disorders) | 22 | 14
Mucosal inflammation (General disorders) | 21 | 89
Oedema peripheral (General disorders) | 73 | 110
Pain (General disorders) | 21 | 26
Pyrexia (General disorders) | 81 | 84
Nasopharyngitis (Infections and infestations) | 43 | 25
Pneumonia (Infections and infestations) | 11 | 29
Sinusitis (Infections and infestations) | 10 | 22
Upper respiratory tract infection (Infections and infestations) | 34 | 26
Urinary tract infection (Infections and infestations) | 24 | 25
Alanine aminotransferase increased (Investigations) | 29 | 30
Aspartate aminotransferase increased (Investigations) | 34 | 33
Blood alkaline phosphatase increased (Investigations) | 29 | 18
Blood cholesterol increased (Investigations) | 8 | 31
Blood creatinine increased (Investigations) | 62 | 61
Platelet count decreased (Investigations) | 11 | 21
Weight decreased (Investigations) | 58 | 67
Decreased appetite (Metabolism and nutrition disorders) | 109 | 145
Hypercalcaemia (Metabolism and nutrition disorders) | 27 | 17
Hypercholesterolaemia (Metabolism and nutrition disorders) | 3 | 38
Hyperglycaemia (Metabolism and nutrition disorders) | 38 | 66
Hyperkalaemia (Metabolism and nutrition disorders) | 27 | 20
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 24 | 77
Hyponatraemia (Metabolism and nutrition disorders) | 27 | 24
Arthralgia (Musculoskeletal and connective tissue disorders) | 120 | 79
Back pain (Musculoskeletal and connective tissue disorders) | 99 | 77
Bone pain (Musculoskeletal and connective tissue disorders) | 19 | 22
Flank pain (Musculoskeletal and connective tissue disorders) | 22 | 18
Muscle spasms (Musculoskeletal and connective tissue disorders) | 23 | 18
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 32 | 22
Myalgia (Musculoskeletal and connective tissue disorders) | 40 | 24
Pain in extremity (Musculoskeletal and connective tissue disorders) | 60 | 45
Dizziness (Nervous system disorders) | 40 | 37
Dysgeusia (Nervous system disorders) | 9 | 40
Headache (Nervous system disorders) | 65 | 66
Taste disorder (Nervous system disorders) | 9 | 21
Anxiety (Psychiatric disorders) | 33 | 25
Depression (Psychiatric disorders) | 25 | 14
Insomnia (Psychiatric disorders) | 40 | 38
Pollakiuria (Renal and urinary disorders) | 21 | 15
Cough (Respiratory, thoracic and mediastinal disorders) | 146 | 152
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 36 | 32
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 101 | 114
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 26 | 28
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 19 | 66
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 22 | 17
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 24 | 15
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 21 | 27
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 13 | 22
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 24 | 56
Productive cough (Respiratory, thoracic and mediastinal disorders) | 23 | 25
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 14 | 24
Dry skin (Skin and subcutaneous tissue disorders) | 50 | 50
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 22 | 38
Pruritus (Skin and subcutaneous tissue disorders) | 92 | 64
Rash (Skin and subcutaneous tissue disorders) | 86 | 101
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 21 | 24
Hypertension (Vascular disorders) | 49 | 47
Hypotension (Vascular disorders) | 24 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.